CLINICAL TRIAL: NCT01417845
Title: The Effect of Moderate Versus High Intensity Exercise Training on Physical Fitness and Physical Function in Patients With Type 2 Diabetes: A Randomized Clinical Trial
Brief Title: The Effect of Exercise Training Intensity in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Arkansas (Other)
Responsible Party: Principal Investigator, James David Taylor, PT, PhD, Associate Professor of Physical Therapy, University of Central Arkansas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCA-IRB-11-077
Record Dates: First submitted 2011-08-11; First posted 2011-08-16 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Intensity Exercise (Experimental): High intensity resistance and aerobic training
  Interventions: Behavioral: High Intensity Exercise Training
- Moderate Intensity Exercise (Active Comparator): Moderate intensity resistance and aerobic training
  Interventions: Behavioral: Moderate Intensity Exercise Training

INTERVENTIONS:
Behavioral: High Intensity Exercise Training — * High intensity resistance and aerobic training
  * Resistance training is performed 2 days per week for 3 months
  * Aerobic training is performed on the same days as resistance training and 1 additional day per week.
  Arms: High Intensity Exercise
Behavioral: Moderate Intensity Exercise Training — * Moderate intensity resistance and aerobic training
  * Resistance training is performed on 2 days per week for 3 months.
  * Aerobic training is performed on the same days as resistance training and 1 additional day per week.
  Arms: Moderate Intensity Exercise

SUMMARY:
The purpose of this randomized clinical trial is to compare the effect of moderate versus high intensity exercise training on physical fitness and physical function in patients with type 2 diabetes. The research hypothesis is that high intensity exercise training will be superior to moderate intensity on such outcomes in individuals with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* All participants meet the American Diabetes Association diagnostic criteria for type 2 diabetes.
* A physician must consider each participant to be medically stable to participate in this investigation.

Exclusion Criteria:

* Any individual with a history of a medical condition identified by the American Heart Association as an absolute contraindication to exercise testing is excluded from this study.
* Any individual with angina (stable or unstable), uncontrolled hypertension, proliferative retinopathy, severe peripheral neuropathy, nephropathy, autonomic neuropathy, history of coronary artery disease, history of myocardial infarction, or unable to participate in this study due to a physical impairment is excluded from this investigation.
* Any individual involved in resistance training or aerobic training within 3 months of the beginning of this investigation is excluded.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-09; Primary Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Muscle Strength | Baseline and 3 months thereafter
Physical Function | Baseline and 3 months thereafter
Exercise Capacity | Baseline and 3 months thereafter

CONTACTS AND LOCATIONS:
Overall Officials: James D Taylor, PhD, PT, Principal Investigator — University of Central Arkansas
Locations (1):
- University of Central Arkansas, Conway, Arkansas, United States

REFERENCES:
- [Derived] Taylor JD, Fletcher JP, Mathis RA, Cade WT. Effects of moderate- versus high-intensity exercise training on physical fitness and physical function in people with type 2 diabetes: a randomized clinical trial. Phys Ther. 2014 Dec;94(12):1720-30. doi: 10.2522/ptj.20140097. Epub 2014 Jul 31. PMID 25082918